CLINICAL TRIAL: NCT06630806
Title: A First-in-human, Open-label, Phase 1 Study to Evaluate the Safety, Antitumor Activity, Pharmacokinetics, and Pharmacodynamics of Subcutaneous SAR446523, an Anti-GPRC5D ADCC-enhanced Monoclonal Antibody, in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Investigate the Safety and Efficacy of SAR446523 Injected Subcutaneously in Adult Participants With Relapsed/Refractory Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED18162; U1111-1301-4016 (Other: WHO ICTRP); 2024-511667-28 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Plasma Cell Myeloma Refractory
Keywords: anti-GPRC5D NK cell targeting therapy

STUDY DESIGN:
Intervention Model Description: Study is non-randomized for part A but randomized for part B. Study drug will be assigned in sequential manner in Part A but parallel assignment in Part B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Dose escalation) (Experimental): Participants will receive SAR446523
  Interventions: Drug: SAR446523
- Part B Dose-1 (Dose optimization) (Experimental): Participants will receive SAR446523 Dose-1
  Interventions: Drug: SAR446523
- Part B Dose-2 (Dose optimization) (Experimental): Participants will receive SAR446523 Dose-2
  Interventions: Drug: SAR446523

INTERVENTIONS:
Drug: SAR446523 — Pharmaceutical form: Powder for solution for injection; Route of administration: Subcutaneous (SC)

SUMMARY:
This is a first-in-human study of SAR446523 conducted in patients with RRMM.

The study consists of two parts:

Dose escalation (Part A): In this part, up to 6 dose levels (DLs) of SAR446523 will be explored to determine the maximum administered dose (MAD), maximum tolerated dose (MTD), and recommended dose range (RDR) of 2 dose regimens which will be tested in the dose optimization part.

Dose optimization (Part B): In this part, participants will be randomly assigned in a 1:1 ratio using interactive response technology (IRT) to either one of the chosen dose regimens of SAR446523 (determined from data coming from Part A), to determine the optimal dose as the recommended phase 2 dose (RP2D) of SAR446523.

DETAILED DESCRIPTION:
The study will be considered ongoing until the last participant last visit has occurred. Participants will be allowed to continue therapy until disease progression, unacceptable AEs, participant or Investigator's request to discontinue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a documented diagnosis of multiple myeloma (MM) with measurable disease.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Dose escalation (Part A)

* Participants must have received at least 3 prior lines of antimyeloma therapy, and must be either relapsed or refractory to the above therapies, or are intolerant to them.
* Note: In Part A, prior exposure to anti g-protein-coupled receptor, class c, group 5, member d (GPRC5D) therapy and anti B-cell maturation antigen (BCMA) therapy is allowed.

Dose optimization (Part B)

* Participants must have received at least 3 prior lines of antimyeloma therapy and be either relapsed or refractory to immunomodulator (IMiD), proteasome inhibitor (PI), anti CD38 monoclonal antibody (mAb), and anti BCMA targeting agent or are intolerant to them.
* Note: In Part B, prior exposure to antiGPRC5D therapy is not allowed.

Exclusion Criteria:

-Participants are excluded from the study if any of the following criteria apply: Eastern cooperative oncology group performance status (ECOG PS) of 2 or greater.

* Primary systemic and localized amyloid light chain (AL) amyloidosis, active polyneuropathy, organomegaly, endocrinopathy, myeloma protein, and skin changes (POEMS) syndrome, active plasma cell leukemia. Participants with central nervous system involvement or with clinical signs of meningeal involvement of multiple myeloma.
* Systemic antimyeloma treatment within 14 days before the first study treatment administration.
* Prior treatment with natural killer (NK)-cell engaging therapy (such as monoclonal antibody with antibody-dependent cellular cytotoxicity as primary mechanism of action) within 90 days of the first study treatment administration.
* Inadequate organ and marrow function.
* Participants with significant concomitant illness.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2028-11-13 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs)- Dose escalation (Part A) | Cycle 1 (28 days)
  The incidence of DLTs will be evaluated using NCI CTCAE version 5.0 criteria.
Overall response rate (ORR) - Dose optimization (Part B) | 24 months after the Last Participant In (LPI)
  ORR is defined as the proportion of participants with sCR, CR, VGPR, and PR assessed as per Investigator according to the 2016 IMWG response criteria.

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs), injection related reactions (IRRs), injection site reactions (ISRs), serious adverse events (SAEs), adverse event of special interests (AESIs) | From the signing of informed consent to 30 days after the date of the last study treatment administration i.e., approximately 5 years
  Measured as per NCI CTCAE v 5.0
Change from baseline in laboratory abnormalities | From the signing of informed consent to 30 days after the date of the last study treatment administration i.e., approximately 5 years
  Measured as per NCI CTCAE v 5.0.
ORR- Dose escalation (Part A) | 24 months after the Last Participant In (LPI)
  ORR defined as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) assessed as per Investigator according to the 2016 International Myeloma Working Group (IMWG) response criteria.
VGPR or better rate | 24 months after the Last Participant In (LPI)
  VGPR or better rate defined as the proportion of participants with sCR, CR, and VGPR assessed as per Investigator according to the 2016 IMWG response criteria.
Clinical benefit rate (CBR) | 24 months after the Last Participant In (LPI)
  CBR defined as the rate of participants with confirmed sCR, CR, VGPR, or PR at any time or minimal response (MR) of at least 6 months from the first IMP administration determined per 2016 IMWG response criteria.
Duration of response (DoR) | 24 months after the Last Participant In (LPI)
  DoR defined as the time from the date of the first response (PR or better) to the date of first documentation of progressive disease (PD) as defined in the 2016 IMWG response criteria, or date of death, whichever occurs first.
Time to response (TTR) | 24 months after the Last Participant In (LPI)
  TTR defined as the time from the first administration of study IMP to the date of first response (PR or better) that is subsequently confirmed.
Progression free survival (PFS) | 24 months after the Last Participant In (LPI)
  PFS defined as the time interval from the date of first administration of study IMP to the date of first documentation of PD per 2016 IMWG criteria assessed by study Investigator, or date of death from any cause, whichever comes first.
Minimal residual disease (MRD) status negativity | 24 months after the Last Participant In (LPI)
  MRD status negative by nextgeneration sequencing (NGS) in bone marrow of participants with a response of CR (or VGPR in case of suspected interference).
Number of participants with symptomatic AEs -Part B | From Cycle 1 Day 1 to 30 days after the date of the last study treatment administration i.e., approximately 5 years
  The incidence and evaluation of symptomatic AEs from participants' perspective will be measured by using specific items from National Cancer Institute (NCI) patient-reported outcome (PRO) common terminology criteria for adverse events (CTCAE) library.
Change from baseline in overall side effect bother as measured by the Functional Assessment of Cancer Therapy item 5 (FACT-GP5)- Part B | From Cycle 1 Day 1 to 30 days after the date of the last study treatment administration i.e., approximately 5 years
  The FACT GP5 is an assessment focused on the overall side effect impact to inform the tolerability of a treatment. The FACT GP5 ("I am bothered by side effects of treatment") responses are given on a 5 point Likert type scale recalling the past 7 days. Higher scores indicate a higher degree of side effect bother.
Maximum observed concentration (Cmax) | Multiple timepoints from Cycle 1 Day 1 to Cycle 1 Day 8 (cycle 1=28 days)
  To characterize the pharmacokinetics (PK) of SAR446523.
First time to reach Cmax (tmax) | Multiple timepoints from Cycle 1 Day 1 to Cycle 1 Day 8 (cycle 1=28 days)
  To characterize the PK of SAR446523.
Area under the concentration versus time curve calculated from 0 to 168 hours (AUC0-168h) | Multiple timepoints from Cycle 1 Day 1 to Cycle 1 Day 8 (cycle 1=28 days)
  To characterize the PK of SAR446523.
Proportion of participants with presence of anti-drug antibody (ADA) against SAR446523. | From Cycle 1 Day 1 to 90 days after the date of the last study treatment administration i.e., approximately 5 years
  To evaluate potential immunogenicity.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (5):
  - Mayo Clinic in Arizona - Phoenix- Site Number : 8400005, Phoenix, Arizona
  - Mayo Clinic in Florida- Site Number : 8400003, Jacksonville, Florida
  - Mayo Clinic in Rochester - Minnesota- Site Number : 8400004, Rochester, Minnesota
  - Hackensack Meridian Health - Hackensack University Medical Center- Site Number : 8400001, Hackensack, New Jersey
  - Thomas Jefferson University Hospital- Site Number : 8400002, Philadelphia, Pennsylvania
- Australia (2):
  - Investigational Site Number : 0360001, Wollongong, New South Wales
  - Investigational Site Number : 0360002, Melbourne, Victoria
- Canada (2):
  - Investigational Site Number : 1240001, Montreal, Quebec
  - Investigational Site Number : 1240002, Sherbrooke, Quebec
- France (2):
  - Investigational Site Number : 2500002, Lille
  - Investigational Site Number : 2500001, Nantes
- Israel (3):
  - Investigational Site Number : 3760001, Tel Aviv, Malopolskie
  - Investigational Site Number : 3760004, Haifa
  - Investigational Site Number : 3760002, Jerusalem
- Italy (2):
  - Investigational Site Number : 3800002, Torette, Ancona
  - Investigational Site Number : 3800001, Rozzano, Milano
- Spain (2):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TED18162 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26146&tenant=MT_SNY_9011